CLINICAL TRIAL: NCT06637735
Title: The Effect of Education Given to Pregnant Women on the Perception of Traumatic Childbirth
Brief Title: The Effect of Education on Pregnant Women Perception of Traumatic Childbirth
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sakarya University (Other)
Responsible Party: Principal Investigator, GÜLESER ADA, Research Asisstant, Sakarya University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SAU-EBE-GA-01
Record Dates: First submitted 2024-09-21; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Pregnant Women; Education
Keywords: education; pregnancy; traumatic childbirth
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: experimental and control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Experimental group; pregnant women will receive a 4-week training
  Interventions: Other: education
- control (No Intervention): No intervention will be made to the control group. Only measurements will be made on parallel dates with the experimental group.

INTERVENTIONS:
Other: education — pregnant women will be given a 4-week training and the pre-test post-test will be analyzed
  Arms: Experimental group

SUMMARY:
During pregnancy, women are exposed to physical, psychological and social changes and may experience anxiety and fears about childbirth. Traumatic birth perception is defined as perceiving birth as a threat to oneself and one's baby. This perception can negatively affect women's lives in the postpartum period. Midwives are the primary health professionals in preventing traumatic birth perception. In this context, it is envisaged to create an important basis for preventing traumatic birth perception in pregnant women through the training to be given.

DETAILED DESCRIPTION:
One of the most important goals of the World Health Organization is to achieve integrated and quality care that creates positive pregnancy and childbirth experiences for women (WHO 2016). Pregnancy is one of the most vulnerable periods in a woman's life and it is possible to predict most of the deaths that occur during pregnancy or childbirth; therefore, providing health care during and after pregnancy is one of the main strategies to improve the health and prevent deaths of mothers and babies (Doaltabadi et al. 2021). In our country, childbirth preparation training has been included in education and practice in different forms for many years. Birth preparation class (DHS) related pieces of training started in the 1990s. Childbirth education classes prepare pregnant women for childbirth and can be done individually or in groups. These courses aim to improve women's lifestyles during pregnancy, birth, and postpartum while protecting infant and maternal rights (Krysa et al., 2016). Education and group interactions allow mothers to share their experiences and knowledge and support each other. Participation in these educational courses includes reducing fear of childbirth and increasing awareness of the potential risks of cesarean section, which leads to improved pregnancy outcomes (Kordi et al. 2017). Studies on the effectiveness of prenatal education have yielded conflicting results. One study showed that this training significantly reduced the fear of childbirth in pregnant women and increased the desire for natural birth (Mousavi et al. 2021). On the other hand, another study did not show a significant effect of this training on reducing anxiety and increasing mothers' self-efficacy (Khaikin et al. 2016). It was also reported that this training reduced labor anxiety but did not affect the duration and mode of labor (Artieta-Pinedo et al. 2010). According to the results of Lee and Holroyd, pregnant women participating in childbirth preparation courses can manage their pregnancy and postpartum better than women who receive only routine care (Lee and Holroyd 2009). When the studies were examined, it was seen that most of the studies were conducted on fear of childbirth and a study on traumatic birth perception has not been found yet. Various health education methods such as face-to-face education, brochures, clips and educational mass media have been used for decades to motivate healthy behaviors in pregnant women.

During pregnancy, expectant mothers often seek information and support to better prepare for birth. Traditionally, pregnant women have relied on books, health professionals, and face-to-face childbirth education classes for information. Given the importance of educating pregnant women about appropriate prenatal care and the potential for education to improve these activities, this study will examine the impact of education on reducing perceptions of traumatic birth in pregnant women.

Place of the study: The study will be conducted with pregnant women admitted to Bartın Maternity and Pediatric Hospital.

Population and sample of the study: The population of the study will consist of pregnant women admitted to Bartın Maternity and Pediatric Hospital who scored at least 53 points on the Traumatic Birth Perception Scale. The minimum traumatic birth perception scale score is 0 and the maximum is 130. Scale total score 0-26 points range is very low, 27-52 points range is low, 53-78 points range is medium, 79-104 points range is high and 105-130 points range is very high traumatic birth perception level (Yalnız et al., 2016). Before starting the study, power analysis was performed with the G*Power 3.1.9.7 program to determine the number of participants in the intervention and control groups (Faul et al., 2013). As a result of the power analysis applied with the G*Power 3.1.9.7 program, the sample size was determined as 26 people in the groups and 52 people in total according to the type 1 error: 0.05 type 2 error: 0.20 and effect size = 0.80 for the determination of the difference between the groups in terms of measurements. Considering the calculated situation due to possible losses in the study, the sample size was increased by 20% and it was planned to take 62 pregnant women, 31 in groups. Pregnant women participating in the study will not be informed which group they are in. Blinding will not be done because the researcher is involved in grouping, intervention and data collection.

Inclusion Criteria:

* Volunteering to participate in the study,
* 18 years of age or older,
* At least 53 points from the Traumatic Birth Perception Scale
* No pregnancy-related risks (such as pre-eclampsia, diabetes, heart disease, placenta previa, oligohydramnios),
* The fetus has no health problems (fetal anomaly, intrauterine growth retardation, etc.),
* Literate,

Exclusion Criteria:

* Refused to participate in the study,
* Illiterate,
* Has a disorder based on a psychiatric/psychological diagnosis,
* Pregnant women with communication and language problems will not be included in the study.

Variables of the Study Independent Variables Information on sociodemographic (age, education, family type, employment status, etc.) and obstetric characteristics (gestational week, gravida, parity, etc.) of pregnant women were the independent variables of the study.

Dependent Variables Traumatic Birth Perception Scale and E-Health Literacy in Pregnant Women Scale constitute the dependent variables.

Data collection tools:

Pregnant Introductory Information Form: This form was developed in line with the literature (Noordam et al., 2011; Lagan et al., 2011; Evans et al., 2012; Parker et al., 2012; Gökçe İsbir & İnci, 2014; Yamin et al., 2016; Yalnız et al., 2016). The study consisted of 8 questions including information about women's sociodemographic (age, education period, family type, employment status) and obstetric characteristics (gestational week, sex of the baby). The Pregnant Introductory Information Form will be completed after the informed consent form and voluntary consent form are completed.

Traumatic Perception of Childbirth Scale: The scale was developed by Yalnız et al. in 2016 to determine the traumatic perception of childbirth. Traumatic perception of birth consists of 13 questions including women's thoughts about the moment of birth. Women's agreement with the given statements was graded between 0 (positive thought) and 10 (negative thought). It is possible to score between 0 and 130 points from the scale. The total mean score of the scale shows that the level of TDA is 0-26 very low, 27-52 low, 53-78 medium, 79-104 high and 105-130 very high. The Cronbach Alpha internal consistency coefficient of the scale was found to be 0.89 (Yalnız, 2016).

E-Health Literacy Scale in Pregnant Women: The scale was developed by Ada and İlçioğlu (2024). The scale consists of 2 sub-dimensions. A minimum score of 1 and a maximum score of 65 is obtained from the scale. There are no reverse coded items in the scale. The scale consists of 13 items. The Cronbach's alpha internal reliability coefficient of the scale was 0.933 and the sub-dimension reliabilities were found to be reliable in the range of 0.910-0.894.

Data Analysis: In the study, the data will be entered into the database in IBM SPSS 26.0 (Statistical Package for the Social Sciences) and AMOS 24 package program and analyzed. While evaluating the study data, frequency distribution (number, percentage) for categorical variables and descriptive statistics (mean, standard deviation, median, minimum, maximum) for numerical variables will be given. The independent sample t-test will be used for the differences between the variables if they conform to the normal distribution, and the Mann Whitney U test will be used if they do not conform to the normal distribution. In addition, in order to examine the change in measurements over time, the dependent sample t test will be used for those who comply with the normal distribution, Wilcoxon test for those who do not comply with the normal distribution and Crombach alpha value for scale reliability. For significance, p<0.05 will be accepted.

Ethics Committee permission was obtained for the implementation of the study. Institutional permission was obtained from Bartın Provincial Health Directorate and Bartın State Hospital before the research.

Each group will consist of pregnant women who scored at least 53 points on the Perception of Traumatic Birth Scale.

A 4-week training will be given online to the Experimental Group. The content of the training will be creaated in line with the expectations of the pregnant women.

The content of the training will be based on Beck's (2015) Traumatic Birth Mid-Range Theory and will be created by aiming to help pregnant women have a healthy pregnancy and birth process with supportive and educational midwifery system recommendations.

Pregnant women included in the groups will be administered the Traumatic Birth Perception Scale and the E-Health Literacy Scale in Pregnant Women as a pre-test. Then, after 4 weeks of training, the post-test will be applied to the pregnant women; Traumatic Birth Perception Scale and E-Health Literacy Scale for Pregnant Women will be applied.

ELIGIBILITY:
Inclusion Criteria: - Volunteering to participate in the study,

* 18 years of age or older,
* At least 53 points from the Traumatic Birth Perception Scale
* No pregnancy-related risks (such as pre-eclampsia, diabetes, heart disease, placenta previa, oligohydramnios),
* The fetus has no health problems (fetal anomaly, intrauterine growth retardation, etc.),
* Literate,

Exclusion Criteria: - Refused to participate in the research,

* Illiterate,
* Has a disorder based on a psychiatric/psychological diagnosis,
* Pregnant women with communication and language problems will not be included in the study.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 62 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
pre-test post-test | 1 month
  The traumatic Childbirth Perception scale in pregnant women will be used as a pre-test and post-test. The experimental and control groups of the study will consist of pregnant women who scored at least 53 points on the Traumatic Childbirth Perception Scale. The minimum traumatic birth perception scale score is 0, and the maximum is 130. Scale total score 0-26 points range is very low, 27-52 points range is low, 53-78 points range is medium, 79-104 points range is high, and 105-130 points range is very high traumatic birth perception level.

CONTACTS AND LOCATIONS:
Overall Officials: Güleser ADA, Master, Study Chair — sakarya üniversity
Locations (1):
- Sakarya Üniversity, Türkiye, Sakarya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No